CLINICAL TRIAL: NCT03481621
Title: Pilot Clinical Trial of Two Acupuncture Protocols on Vulvodynia
Brief Title: Effect of Two Acupuncture Protocols on Vulvodynia
Acronym: Acu/Vul-pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: McLean Center for Complementary and Alternative Medicine, PLC (Other)
Responsible Party: Principal Investigator, Arthur Fan, Director,Principal Investigator, McLean Center for Complementary and Alternative Medicine, PLC
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: McLeanCCAM01
Record Dates: First submitted 2018-03-08; First posted 2018-03-29 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-09

CONDITIONS: Vulvodynia; Vulvodynia, Generalized; Vulvar Vestibulitis; Vulvar Pain
Keywords: Vulvodynia
MeSH Terms: conditions — Vulvodynia; Vulvar Vestibulitis | interventions — Acupuncture Therapy; Standard of Care

STUDY DESIGN:
Intervention Model Description: Acupuncture 1: focus on the points within pudendal nerve distribution arae; Acupuncture 2: focus on the points from traditional meridian theory; Standard care: no acupuncture, but use physical therapy, pain medications, nerve blocking, etc.
Who Masked: Participant, Outcomes Assessor
Masking Description: All participants will get real treatments, the first group patients will get acupuncture treatments focus on the points within pudendal nerve distribution area; the second group patients will get acupuncture treatments focus on the points from traditional meridian theory. And the third group will get the standard care (no acupuncture). Participants and outcomes assessor will be blinded for the study aims.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Group1a, Acupuncture on Vulvodynia (Active Comparator): Focus on using the local points in pudendal nerve distribution area
  Interventions: Device: Acupuncture
- Group1b, Acupuncture on Vulvodynia (Active Comparator): Focus on traditional acupuncture using common meridian or distal points
  Interventions: Device: Acupuncture
- Group2, Standard care or waiting lists (Active Comparator): Standard care without acupuncture
  Interventions: Other: Standard care

INTERVENTIONS:
Device: Acupuncture — Needle size: #32(0.22 mm), 1-1.5 inch(30-40 mm long); Acupuncture time and frequency: 45 min per session, once or twice per week, for 6-12 sessions total (in 6 weeks).
  Other Names: Needling
  Arms: Group1a, Acupuncture on Vulvodynia; Group1b, Acupuncture on Vulvodynia
Other: Standard care — PT, pain medications, nerve block, etc
  Other Names: Routine treatments
  Arms: Group2, Standard care or waiting lists

SUMMARY:
Vulvodynia is a common condition in women (16%); however, at this time there is no known effective non-pharmacological therapy reported. Acupuncture is one complementary and alternative medicine therapy used by many patients with vulvodynia; some case reports show that acupuncture may be an effective intervention. In recent years, there were some studies registered took at like at actual trials of acupuncture on vulvodynia, but either they did not reach the trial aims, some studies did not get enough patients or the trial designs mimic drug studies and did not reflect acupuncture real characteristics.

This study evaluates acupuncture for the treatment of vulvodynia; specifically, if it reduces vulvar pain, pain duration and pain with intercourse. It also examines how long the effect of acupuncture lasts in women with vulvodynia. One third of the women will receive acupuncture focused on pudendal nerve distribution area; another one third of the women will receive acupuncture focused on traditional meridian points; the other one third of women will use standard care (without acupuncture). Women who get a reduction in pain (included in subjective and objective scores) will have their pain monitored once a week for up to 6 weeks to see if the acupuncture effect lasts.

DETAILED DESCRIPTION:
Aims of this study:

1. Get preliminary data for future larger, randomized- controlled trials.
2. See whether acupuncture is better than no-acupuncture treatments (where participations are following standard care for this condition), or at least have probable better outcomes than no acupuncture treatment (there may not be significance in statistics, given the small sample in current proposed trial);
3. See if acupuncture group 1a (with focus on the points in pudendal nerve distribution near the pain area) has better results(at least, a trend) than acupuncture group 1b (traditional acupuncture focus on meridian or distal points).

The basic design and interventions:

1. Diagnosis: Vulvodynia/Vulval pain by gynecologist or pain specialist/doctor, who will adopt International diagnose criteria.
2. Patient sample (estimated): 17 in each acupuncture group (34 total), and 17 patients in the no-acupuncture group or standard care waiting list . Total 51 patients;
3. Groups:

   Group 1a (17 cases): acupuncture, using the local points in pudendal nerve distribution area (tender points, and up to two other set of acupuncture points); Group 1b (17 cases): traditional acupuncture, using common meridian or distal points; Group 2 (17 cases): standard care, waiting list. This group will receive no acupuncture treatment.
4. Randomized method: If the patient feels comfortable with acupuncture, they will be randomly assigned to either Group 1a or Group1b using randomization numbers generated by computer; if the patients still are under the treatments of routine conventional treatments, such as using pain medications, local injections, and physical therapies, or other non-surgical procedure, they will serve as participants in the standard care group, the waiting list.
5. Blind Method: Patients will be blind as to the purpose of the study as well as to the groups that they are assigned too. Each participant in either group 1a or 1b will receive actual, real acupuncture treatment but, depending on their group assignment, the strategy and points used will vary.
6. Treatments:

   Group 1a: acupuncture: needling focus on Hui yang, pudendal nerve points and local point(s) near the pain location with needling manipulation (such as twisting 200/min for 2-5 minutes at pudendal nerve points); Group 1b: acupuncture: using meridian points, focus on Xue Hai (SP9), San Yin Jiao (SP6), Zu San Li (ST36); Both groups also use: Shen Ting (GV24), Tou Wei (ST 8), Yin Tang (EX2) for helping to release stress and create calm.

   Both group 1(a/b) and group 2 patients are all allowed to use pain medications (in which the medications' name and how many pills used during 6 weeks' observation period will be carefully document); the standard care group actually is a waiting list, without acupuncture intervention. Follow up: 6 weeks.

   Acupuncture time and frequency: 45 min per session, once or twice per week, for 6-12 sessions (in 6 weeks).
7. Main observation:

(1) Objective pain score(tested using cotton swab); (2) Patient self reported pain score (subjective, before Cotton swab test); Others: Pain duration and pain score during intercourse.

8. Statistics: student t-test.

Sample calculation: The expected difference (ECSD) between two means is 3, and the common within group standard deviation is 3. Giving an 80 chance that an 0.05 level test of significance will find a statistically significant difference between two sample means are compared, the sample size is approximately 17 per group.

Comparisons:

1. At the end point (end of 6 weeks), make comparisons between acupuncture (1a+1b) group and group 2, acupuncture 1a and group 2, acupuncture 1b and group 2; between acupuncture 1a and acupuncture 1b; respectively.
2. At the end point (end of 6 weeks), make comparisons in each group self (before and after).

ELIGIBILITY:
Inclusion Criteria:

1. diagnosis of generalized vulvodynia or provoked vestibulodynia by OB/GYN doctor(s) or pain specialist(s); 18 to 45 years old.
2. Current pain score 4 or higher with tampon insertion and removal performed, or cotton swab test, at the initial screening exam
3. speak and read English or Chinese.

Exclusion Criteria:

1. infectious conditions of the vulvar/vagina;
2. inflammatory conditions of the vulvar/vagina;
3. neoplastic disorders of the vulvar/vagina;
4. neurologic disorders of the vulvar/vagina;
5. acute trauma to the genitals;
6. iatrogenic conditions of the genitals
7. hormonal deficiencies
8. co-morbid pelvic pain conditions (to avoid confounding pain outcomes) such as pelvic inflammatory disease and documented history of endometriosis
9. menopause
10. patients have active migraine headaches, temporomandibular joint disease (TMJ), irritable bowel syndrome (IBS), interstitial cystitis, painful bladder syndrome, or fibromyalgia, in past 6 month.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 51 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain Score (objective) | at the end of 6 weeks
  Figure out the pain score using Visual Analog pain scale(VAS) using cotton swab , [score 0-no pain, 10-strongest (unbearable) pain]. Expected clinical significant difference (ECSD): 3.

SECONDARY OUTCOMES:
Pain Score (Subjective) | at the end of 6 weeks
  Figure out the pain score using Visual Analog pain scale(VAS) before use of cotton swab to to test pain , [score 0-no pain, 10-strongest (unbearable) pain]. Expected clinical significant difference (ECSD): 3.
Pain duration | at the end of 6 weeks
  Monitor the hours of pain per day
Intercourse pain | at the end of 6 weeks
  Record how much pain during intercourse using Visual Analog pain scale(VAS) [score 0-no pain, 10-strongest]

CONTACTS AND LOCATIONS:
Overall Officials: Arthur Y Fan, MD(CHN),PhD, Principal Investigator — McLean Center for Complementary and Alternative Medicine, PLC
Locations (1):
- McLean Center for Complementary and Alternative Medicine,PLC, Vienna, Virginia, United States

REFERENCES:
- [Derived] Fan AY, Alemi SF, Zhu YH, Rahimi S, Wei H, Tian H, He D, Gong C, Yang G, He C, Ouyang H. Effectiveness of two different acupuncture strategies in patients with vulvodynia: Study protocol for a pilot pragmatic controlled trial. J Integr Med. 2018 Nov;16(6):384-389. doi: 10.1016/j.joim.2018.10.004. Epub 2018 Oct 10. PMID 30341023